CLINICAL TRIAL: NCT06808568
Title: Expanded Access Program (EAP) STIMULAN VG
Acronym: EAPSTIMVG
Status: Available | Type: Expanded Access
Sponsor: Biocomposites Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EAPSTIMVG
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Stage IV Pressure Ulcer; Diabetic Foot Osteomyelitis
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Combination Product: STIMULAN VG

SUMMARY:
Individual (single) patient expanded access may be considered.

DETAILED DESCRIPTION:
Patients facing serious or life-threatening illnesses who have exhausted currently available treatment options and are ineligible or unable to participate in a clinical trial may decide to explore therapeutic use of investigational drugs with their healthcare providers.

Under these circumstances, single-patient access can be requested from a licensed treating physician on behalf of the patient.

Please contact expandedaccess@biocomposites.com for more information.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult